CLINICAL TRIAL: NCT06122194
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED, SINGLE DOSE, CROSSOVER STUDY TO ESTIMATE THE RELATIVE BIOAVAILABILITY OF PF-07817883 FOLLOWING ORAL ADMINISTRATION OF NEW FORMULATIONS RELATIVE TO THE REFERENCE FORMULATION IN HEALTHY ADULT PARTICIPANTS UNDER FASTED CONDITION
Brief Title: A Study to Learn PF-07817883 Blood Levels After Administration of Tablets of Study Drug to Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: C5091013; 2023-506442-24-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-10-10; First posted 2023-11-08 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-09

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: 4 period 4 sequence crossover design
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Period 1 formulation 1 PF-07817883 (Experimental): Single oral dose of PF-07817883 tablet under fasted condition
  Interventions: Drug: Drug: PF-07817883
- Period 2 formulation 2 PF-07817883 (Experimental): Single oral dose of PF-07817883 tablet under fasted condition
  Interventions: Drug: Drug: PF-07817883
- Period 3 formulation 3 PF-07817883 (Experimental): Single oral dose of PF-07817883 tablet under fasted condition
  Interventions: Drug: Drug: PF-07817883
- Period 4 formulation 4 PF-07817883 (Experimental): Single oral dose of PF-07817883 tablet under fasted condition
  Interventions: Drug: Drug: PF-07817883

INTERVENTIONS:
Drug: Drug: PF-07817883 — PF-07817883 tablet

SUMMARY:
The purpose of this study is to estimate the oral bioavailability of 3 new formulations of PF-07817883 (test) relative to reference tablet formulation in healthy adult participants under fasted conditions. The study will also assess the safety and tolerability of test and reference tablet formulations in healthy adult participants.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, randomized, 4-period, 4-sequence crossover study in healthy adult participants evaluating the rBA of 3 new PF-07817883 test oral formulation(s) compared to PF-07817883 reference oral formulation. Approximately 12 participants will be enrolled in this study with approximately equal number of participants randomized to 1 of 4 sequences.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 18 years or older, at screening who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and standard 12-lead ECG.
* BMI of 16 to 32 kg/m2; and a total body weight >45 kg
* Capable of giving signed informed consent.

Exclusion Criteria:

* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior, laboratory abnormality, or other conditions and situations that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).

  1. Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
  2. History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, or HCVAb. Hepatitis B vaccination is allowed.
* Positive test result for SARS-CoV-2 infection at admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5091013

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 12 participants were enrolled and randomized in this study to 1 of the 4 study treatment sequences.
Groups:
- Treatment Sequence 1: A Then B Then C Then D: Participants were randomized to receive a single oral dose of treatment A on Day 1 of Period 1; followed by a single oral dose of treatment B on Day 1 of Period 2; followed by a single oral dose of treatment C on Day 1 of Period 3; followed by a single oral dose of treatment D on Day 1 of Period 4. Between 2 doses of consecutive period there was a gap of at least 48 hours (2 days). A=PF-07817883 300 milligram (mg) tablet reference formulation, B=PF-07817883 300 mg tablet test formulation 1, C=PF-07817883 300 mg tablet test formulation 2 and D=PF-07817883 300 mg tablet test formulation 3. All formulations were administered under fasting condition.
- Treatment Sequence 2: B Then D Then A Then C: Participants were randomized to receive a single oral dose of treatment B on Day 1 of Period 1; followed by a single oral dose of treatment D on Day 1 of Period 2; followed by a single oral dose of treatment A on Day 1 of Period 3; followed by a single oral dose of treatment C on Day 1 of Period 4. Between 2 doses of consecutive period there was a gap of at least 48 hours (2 days). A=PF-07817883 300 mg tablet reference formulation, B=PF-07817883 300 mg tablet test formulation 1, C=PF-07817883 300 mg tablet test formulation 2 and D=PF-07817883 300 mg tablet test formulation 3. All formulations were administered under fasting condition.
- Treatment Sequence 3: C Then A Then D Then B: Participants were randomized to receive a single oral dose of treatment C on Day 1 of Period 1; followed by a single oral dose of treatment A on Day 1 of Period 2; followed by a single oral dose of treatment D on Day 1 of Period 3; followed by a single oral dose of treatment B on Day 1 of Period 4. Between 2 doses of consecutive period there was a gap of at least 48 hours (2 days). A=PF-07817883 300 mg tablet reference formulation, B=PF-07817883 300 mg tablet test formulation 1, C=PF-07817883 300 mg tablet test formulation 2 and D=PF-07817883 300 mg tablet test formulation 3. All formulations were administered under fasting condition.
- Treatment Sequence 4: D Then C Then B Then A: Participants were randomized to receive a single oral dose of treatment D on Day 1 of Period 1; followed by a single oral dose of treatment C on Day 1 of Period 2; followed by a single oral dose of treatment B on Day 1 of Period 3; followed by a single oral dose of treatment A on Day 1 of Period 4. Between 2 doses of consecutive period there was a gap of at least 48 hours (2 days). A=PF-07817883 300 mg tablet reference formulation, B=PF-07817883 300 mg tablet test formulation 1, C=PF-07817883 300 mg tablet test formulation 2 and D=PF-07817883 300 mg tablet test formulation 3. All formulations were administered under fasting condition.
Period: Treatment Period 1 (3 Days)
Arm/Group | Treatment Sequence 1: A Then B Then C Then D | Treatment Sequence 2: B Then D Then A Then C | Treatment Sequence 3: C Then A Then D Then B | Treatment Sequence 4: D Then C Then B Then A
Started | 3 | 3 | 3 | 3
Treated | 3 | 3 | 3 | 3
Completed | 3 | 3 | 2 | 3
Not Completed | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Period: Treatment Period 2 (3 Days)
Arm/Group | Treatment Sequence 1: A Then B Then C Then D | Treatment Sequence 2: B Then D Then A Then C | Treatment Sequence 3: C Then A Then D Then B | Treatment Sequence 4: D Then C Then B Then A
Started | 3 | 3 | 2 | 3
Completed | 3 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 3 (3 Days)
Arm/Group | Treatment Sequence 1: A Then B Then C Then D | Treatment Sequence 2: B Then D Then A Then C | Treatment Sequence 3: C Then A Then D Then B | Treatment Sequence 4: D Then C Then B Then A
Started | 3 | 3 | 2 | 3
Completed | 3 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 4 (3 Days)
Arm/Group | Treatment Sequence 1: A Then B Then C Then D | Treatment Sequence 2: B Then D Then A Then C | Treatment Sequence 3: C Then A Then D Then B | Treatment Sequence 4: D Then C Then B Then A
Started | 3 | 3 | 2 | 3
Completed | 3 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants randomly assigned to study treatment and who took at least 1 dose of study treatment in at least one treatment period. Participants were analyzed according to the product they actually received.
Groups:
- Treatment Sequence 1: A Then B Then C Then D: Participants were randomized to receive a single oral dose of treatment A on Day 1 of Period 1; followed by a single oral dose of treatment B on Day 1 of Period 2; followed by a single oral dose of treatment C on Day 1 of Period 3; followed by a single oral dose of treatment D on Day 1 of Period 4. Between 2 doses of consecutive period there was a gap of at least 48 hours (2 days). A=PF-07817883 300 mg tablet reference formulation, B=PF-07817883 300 mg tablet test formulation 1, C=PF-07817883 300 mg tablet test formulation 2 and D=PF-07817883 300 mg tablet test formulation 3. All formulations were administered under fasting condition.
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence 1: A Then B Then C Then D | Treatment Sequence 2: B Then D Then A Then C | Treatment Sequence 3: C Then A Then D Then B | Treatment Sequence 4: D Then C Then B Then A | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Mean (SD) | 58.7 (4.93) | 34.7 (3.06) | 41.3 (18.15) | 51.0 (21.28) | 46.4 (15.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 1 | 3
  Male | 2 | 2 | 3 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 3 | 2 | 3 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 3 | 3 | 12
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-07817883
Time Frame: 0, 0.5, 1, 2, 4, 6, 8, 12, 24, 48 hours post-dose on Day 1 of each treatment period
Population: Pharmacokinetic (PK) parameter analysis population was defined as all participants randomized and treated who had at least 1 of the PK parameters of interest in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Treatment A: PF-07817883 300 mg Reference Formulation: Participants received PF-07817883 300 mg, tablet, orally as single dose of reference formulation on Day 1 of any period.
- Treatment B: PF-07817883 300 mg Test Formulation 1: Participants received PF-07817883 300 mg, tablet, orally as single dose of test formulation 1 on Day 1 of any period.
- Treatment C: PF-07817883 300 mg Test Formulation 2: Participants received PF-07817883 300 mg, tablet, orally as single dose of test formulation 2 on Day 1 of any period.
- Treatment D: PF-07817883 300 mg Test Formulation 3: Participants received PF-07817883 300 mg, tablet, orally as single dose of test formulation 3 on Day 1 of any period.
Arm/Group | Treatment A: PF-07817883 300 mg Reference Formulation | Treatment B: PF-07817883 300 mg Test Formulation 1 | Treatment C: PF-07817883 300 mg Test Formulation 2 | Treatment D: PF-07817883 300 mg Test Formulation 3
Number analyzed (Participants) | 11 | 11 | 12 | 11
nanogram per milliliter (ng/mL) | 2308 (39) | 2579 (28) | 4266 (40) | 3566 (34)
Statistical Analysis 1: Comparison: Treatment A: PF-07817883 300 mg Reference Formulation vs Treatment B: PF-07817883 300 mg Test Formulation 1; Natural log transformed Cmax for PF-07817883 were analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect in Periods 1 to 4. The ratio (Test/Reference) and 90 percent (%) confidence intervals (CIs) were expressed as percentages; Test type: Other; Ratio of Adjusted Geometric Means = 112.15, 90% CI 2-sided [93.01 to 135.22]
Statistical Analysis 2: Comparison: Treatment A: PF-07817883 300 mg Reference Formulation vs Treatment C: PF-07817883 300 mg Test Formulation 2; Natural log transformed Cmax for PF-07817883 were analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect in Periods 1 to 4. The ratio (Test/Reference) and 90% CIs were expressed as percentages; Test type: Other; Ratio of Adjusted Geometric Means = 187.37, 90% CI 2-sided [155.79 to 225.35]
Statistical Analysis 3: Comparison: Treatment A: PF-07817883 300 mg Reference Formulation vs Treatment D: PF-07817883 300 mg Test Formulation 3; [analysis description as in outcome 1, analysis 2]; Test type: Other; Ratio of Adjusted Geometric Means = 153.61, 90% CI 2-sided [127.40 to 185.21]

2. Primary Outcome: Area Under the Concentration-time Curve From Time Zero (0) Extrapolated to Infinity (AUCinf) of PF-07817883
Time Frame: 0, 0.5, 1, 2, 4, 6, 8, 12, 24, 48 hours post-dose on Day 1 of each treatment period
Population: PK parameter analysis population was defined as all participants randomized and treated who had at least 1 of the PK parameters of interest in at least 1 treatment period. Here, "Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Treatment A: PF-07817883 300 mg Reference Formulation | Treatment B: PF-07817883 300 mg Test Formulation 1 | Treatment C: PF-07817883 300 mg Test Formulation 2 | Treatment D: PF-07817883 300 mg Test Formulation 3
Number analyzed (Participants) | 10 | 9 | 10 | 10
nanogram*hour per milliliter (ng*hr/mL) | 17660 (35) | 18200 (22) | 21040 (36) | 21510 (33)
Statistical Analysis 1: Comparison: Treatment A: PF-07817883 300 mg Reference Formulation vs Treatment B: PF-07817883 300 mg Test Formulation 1; Natural log transformed AUCinf for PF-07817883 were analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect in Periods 1 to 4. The ratio (Test/Reference) and 90% CIs were expressed as percentages; Test type: Other; Ratio of Adjusted Geometric Means = 102.59, 90% CI 2-sided [91.09 to 115.54]
Statistical Analysis 2: Comparison: Treatment A: PF-07817883 300 mg Reference Formulation vs Treatment C: PF-07817883 300 mg Test Formulation 2; [analysis description as in outcome 2, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 125.07, 90% CI 2-sided [110.81 to 141.17]
Statistical Analysis 3: Comparison: Treatment A: PF-07817883 300 mg Reference Formulation vs Treatment D: PF-07817883 300 mg Test Formulation 3; [analysis description as in outcome 2, analysis 1]; Test type: Other; Ratio of Adjusted Geometric Means = 121.75, 90% CI 2-sided [108.65 to 136.43]

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant temporally associated with the use of study treatment, whether or not considered related to the study treatment. Treatment-emergent are events between first dose of study treatment and up to 28-35 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From start of study treatment (Day 1) up to 28-35 days after last dose of study treatment (maximum up to 47 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: PF-07817883 300 mg Reference Formulation | Treatment B: PF-07817883 300 mg Test Formulation 1 | Treatment C: PF-07817883 300 mg Test Formulation 2 | Treatment D: PF-07817883 300 mg Test Formulation 3
Number analyzed (Participants) | 11 | 11 | 12 | 11
Participants | 2 | 2 | 3 | 2

4. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Laboratory parameters included hematology (eosinophils/leukocytes [%] greater than [>] 1.2*upper limit of normal), and urinalysis (urine hemoglobin and leukocyte esterase greater than or equal [>=] to 1).
Time Frame: From start of study treatment (Day 1) up to last dose of study treatment (maximum up to 12 days)
Population: Safety analysis set included all participants randomly assigned to study treatment and who took at least 1 dose of study treatment in at least one treatment period. Participants were analyzed according to the product they actually received. Here, "Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: PF-07817883 300 mg Reference Formulation | Treatment B: PF-07817883 300 mg Test Formulation 1 | Treatment C: PF-07817883 300 mg Test Formulation 2 | Treatment D: PF-07817883 300 mg Test Formulation 3
Number analyzed (Participants) | 3 | 1 | 1 | 3
Participants | 1 | 0 | 1 | 2

5. Secondary Outcome: Number of Participants With Clinically Significant Abnormality in Vital Signs
Description: Vital signs included diastolic blood pressure (DBP), systolic blood pressure (SBP) and pulse rate (PR) were measured in a supine position after approximately 5 minutes of rest for the participant. Criteria for vital signs included: SBP: value less than (<) 90 millimeters of mercury (mmHg), change from baseline greater than or equal to (>=) 30 mmHg increase, change from baseline >=30 mmHg decrease; DBP: value <50 mmHg, change from baseline >=20 mmHg increase, change from baseline >=20 mmHg decrease; PR: value <40 beats per minute (bpm), value greater than (>) 120 bpm.
Time Frame: From start of study treatment (Day 1) up to last dose of study treatment (maximum up to 12 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: PF-07817883 300 mg Reference Formulation | Treatment B: PF-07817883 300 mg Test Formulation 1 | Treatment C: PF-07817883 300 mg Test Formulation 2 | Treatment D: PF-07817883 300 mg Test Formulation 3
Number analyzed (Participants) | 11 | 11 | 12 | 11
Participants | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Clinically Significant Abnormality in Electrocardiogram (ECG)
Description: Standard 12 lead ECGs were obtained with the participant in a supine position after at least 5 minutes of rest. Criteria were PR interval (>=300 millisecond [msec], percent [%] change from baseline >=25 to 50%), QRS duration (>=140 msec, %change from baseline >=50%), corrected QT interval using Fridericia's formula (QTcF) (>500 msec, %change from baseline >60 msec, 450 msec<value less than equal to [<=] 480 msec, 480 msec<value<=500 msec, 30 msec<=change<=60 msec).
Time Frame: From start of study treatment (Day 1) up to last dose of study treatment (maximum up to 12 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: PF-07817883 300 mg Reference Formulation | Treatment B: PF-07817883 300 mg Test Formulation 1 | Treatment C: PF-07817883 300 mg Test Formulation 2 | Treatment D: PF-07817883 300 mg Test Formulation 3
Number analyzed (Participants) | 11 | 11 | 12 | 11
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study treatment (Day 1) up to 28-35 days after last dose of study treatment (maximum up to 47 days)
Description: Safety population included all participants randomly assigned to study treatment, who took at least 1 dose of study treatment. Participants were analyzed according to the product they actually received.
Arm/Group | Treatment A: PF-07817883 300 mg Reference Formulation | Treatment B: PF-07817883 300 mg Test Formulation 1 | Treatment C: PF-07817883 300 mg Test Formulation 2 | Treatment D: PF-07817883 300 mg Test Formulation 3
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 2/11 | 2/11 | 3/12 | 2/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: PF-07817883 300 mg Reference Formulation (N=11) | Treatment B: PF-07817883 300 mg Test Formulation 1 (N=11) | Treatment C: PF-07817883 300 mg Test Formulation 2 (N=12) | Treatment D: PF-07817883 300 mg Test Formulation 3 (N=11)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vessel puncture site bruise (General disorders) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 1
Polyuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-08-24): https://cdn.clinicaltrials.gov/large-docs/94/NCT06122194/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-22): https://cdn.clinicaltrials.gov/large-docs/94/NCT06122194/SAP_001.pdf